CLINICAL TRIAL: NCT01889407
Title: Idarubicin Overcomes Multidrug Resistant-1(MDR1) Induced Chemoresistance With Higher Induction Remission Rate and Remission Quality Than Daunorubicin in de Novo Acute Myeloid Leukemia Patients
Brief Title: Idarubicin Overcomes MDR1 Induced Chemoresistance With Higher Induction Remission Rate and Quality Than Daunorubicin in Acute Myeloid Leukemia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IDA20130517; IDA20130517 (Other: Company of Pfizer)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2013-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Bone marrow
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IA regimen: IA regimen: Patients receive idarubicin (8mg/m2.d) iv drip on days 1-3 and cytarabine (100-200mg/ m2.d) iv drip on days 1-7.
  Interventions: Drug: Idarubicin
- DA regimen: Patients receive daunomycin (45mg/ m2.d) iv drip on days 1-3 and cytarabine (100-200mg/ m2.d) iv drip on days 1-7.

INTERVENTIONS:
Drug: Idarubicin — 8 mg/m2, iv drip on days 1-3
  Groups: IA regimen

SUMMARY:
Whether Idarubicin can overcomes multidrug resistant 1 induced chemoresistance with higher induction remission rate than daunorubicin in de novo acute myeloid leukemia patients.Whether induction therapy with IA regimen has a higher remission quality with AML patients than that of DA regimen in high MDR1 expression AML patients.

DETAILED DESCRIPTION:
The long-term survival rate of acute myeloid leukemia (AML) has been significantly prolonged due to the improvement of chemotherapeutic protocols and hemopoietic stem cell transplantation. However, about 20%-40% of the patients with refractory AML fail to achieve complete remission (CR) and approximately 50% of the CR patients will relapse eventually. 1-3 The refractoried and relapsed AML patients have very poor prognosis, therefore refractoriness and relapse are the major challenges for the chemotherapy of AML.

Chemoresistance is one of the major obstacle for the success of AML treatment.4 One of the main mediators for AML chemoresistance is the multi-drug resistance-1(MDR1) gene and MDR1 protein, also known as permeability-glycoprotein or P-gp.5,6,7 Studies on leukemic blast cells demonstrated the association of MDR1 expression with a lower intracellular retention of cytostatic drugs leading to cancer cell resistance to several commonly used anti-cancer drugs in chemotherapy. Several subsequent studies indicated the influence of MDR1 expression levels in the treatment response and survival of leukemia patients, the frequency of resistance to the chemotherapy increased with increasing MDR1 expression.8,9,10 Previous methods for determination of MDR1 expression have included demonstration of P-glycoprotein by flow cytometry and/or immunohistochemistry, and molecular polymerase chain reaction (PCR)-based assays for RNA expression. However, these assays have either proven difficult to standardize or tedious to perform and they are mainly focused on qualitative or semi-quantitative assays. 11,12 A real-time fluorescence quantitative PCR will increase the sensitivity and also maintain the high specificity. The false positivity caused by pollution of amplification production can also be decreased by hermetization operation. RQ- PCR is a novel methodology which enables sensitive and quantitative measurement of gene expression. 12We have established RQ-PCR method for determination expression of MDR1 gene. We have performed a pilot study with a small cohort of AML patients to determine the relationship of MDR1 expression and CR rate of AML patients. The data shows MDR1 expression has been found in most cases of AML. However, the MDR1 expression levels vary widely from case to case. This result indicated that RQ-PCR method would provide an accurate quantitative measurement for detection of MDR1 expression level in different AML cases who were both positive by qualitative RT-PCR method. 13,14 The pilot results indicated that the complete response rate to induction therapy was compromised by the expression of high levels of MDR1. 15

Minimal residual disease (MRD) is the major cause of leukemia relapse. It has been reported that the treatment intensity in human leukemia can be assessed by the expression status of MRD gene. However, more than 50% of acute leukemia, especially in AMLs, lack known genetic lesions or clonegenic markers suitable for MRD monitoring. WT1 gene is located on chromosome 11p13 coding for a zinc-finger transcription factor, has been identified in most AML patients. It has been reported that detection of WT1 levels can effectively monitor the MRD expression status in AML.16,17 Therefore, WT1 expression can be used to monitor the MRD and evaluation the remission quality in AML patients. By detecting WT1 levels we can evaluate the efficacy of different induction therapies.

By employing multiple fluorescence quantitative PCR, several target genes can be simultaneously and quantitatively amplified. Therefore multiple fluorescence quantitative PCR is more suitable for clinical application. This technology will not only provide higher accuracy, specificity and reproducibility but also simplify procedure and reduce measurement cost. The recombinant plasmids of MDR1 and WT1 gene have been constructed and the methodology of multiple fluorescence quantitative PCR has also been developed in our group .14

High MDR1 gene expression is a common feature of AML resistance to conventional chemotherapeutic regimen.18,19 One of the strategies that overcome MDR is to increase the pharmacal liposolubility and elevate the intracellular drug concentration, so as to counteract drug efflux pumped by P-glycoprotein. Idarubicin (IDA), a new anthracycline, has more strengthened liposolubility and can easily permeate the cell membrane in comparison with traditional marcellomycin. Also, the in vivo metabolite of IDA (4-IDA) has the same antineoplastic activity as IDA and a longer half-life in vivo. It can also permeate blood brain barrier. As a result, IDA has a stronger antileukemia activity than other marcellomycin and can partially overcome P-glycoprotein-mediated drug resistance.20, 21 In our recently pilot study, we have detected the expression of MDR1 in pre-treated bone marrow samples from 160 de novo AML patients and the median value of MDR1/GAPDH ratio in the de novo AML cases was 0.016（0-81.865）. The median value of MDR1 gene expression was taken as the cut-off point of high or low MDR1 gene expression levels. For high MDR1 expression patients, a lower CR rate (61.3%) was observed compared with low-MDR1 expression patients (80.0%, P =0.009). In this retrospective pilot study, 123 patients were received daunorubicin (DNR 35~45mg/m2/d,3 days) or idarubicin (IDA 6~8 mg/m2/d, 3 days) in combination with cytarabine (Ara-c100~200 mg/m2/d, 7 days) for remission induction and significant difference were also observed after 2 courses of chemotherapy between those who receive IA regimen (57 cases) and DA regimen (66 cases) regarding to CR rate (80.7% vs 57.6%, P=0.006). Significant difference could also be discovered between two treatment arm with regard to CR rate (75.9% vs 43.6%, P=0.011) in those who had high MDR1 expression AML patients. Our data shows that IDA may overcome MDR1 induced chemoresistance with a higher CR rate than DNR in de novo high MDR1 expresser AML patients.These results provide rationale for development of randomized, prospective trial to compare the CR rate of IA regimen and DA regimen in de novo AML patients with high MDR1 expression and to identify whether Idarubicin can overcomes MDR1 induced chemoresistance with higher induction remission rate than daunorubicin in de novo acute myeloid leukemia patients. We speculated that the more favorable outcome in high-MDR1 patient group with IA regimen may be associated with a higher remission rate.

It had been reported that AML patients achieved lower MRD level had an extremely lower relapse rate. It had also been reported that patients treated with IA regimen had a significant higher long-term survival than those with DA regimen .22-24 Therefore, we speculated that the more favorable outcome in IA group may be associated with a lower MRD level and higher remission quality. This study is also to conduct a prospective analysis on the alteration of WT1 and MDR1 gene expression level after induction therapy with IA or DA separately to identify whether induction therapy with IA regimen has a lower MRD level and a higher remission quality than that of DA regimen.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of AML (WHO classification definition of >/= 20% blasts).

  * Patients aged 16 to 60 years are eligible. Patients must be chemo-naïve, i.e. not have received any prior chemotherapy (except hydrea) for AML. They could have received transfusion, hematopoietic growth factors or vitamins. Temporary measures such as pheresis or hydrea (0.5 to 5g daily or more for up to 3 days) are allowed.
  * The relative expression level of MDR1 mRNA (MDR1/GAPDH ratio using the quantitative real-time PCR) in pre-treated bone marrow samples should over 0.016 (cut-off point from our results of preliminary experiment data )
  * ECOG PS of 0, 1, 2 at screening.
  * Serum biochemical values with the following limits: - creatinine </= 2.0 mg/dl - total bilirubin </= 2.0 mg/dL, unless increase is due to hemolysis - transaminases (SG PT) </= 3x ULN
  * Ability to understand and provide signed informed consent.

Exclusion Criteria:

* • Subjects with Acute Promyelocytic Leukemia (APL).

  * Presence of active systemic infection.
  * Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results.
  * Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, IUD, diaphragm, abstinence, or condoms by their partner) over the entire course of the study.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: • Patients aged 16 to 60 years are eligible. Patients must be chemo-naïve, i.e. not have received any prior chemotherapy (except hydrea) for AML. They could have received transfusion, hematopoietic growth factors or vitamins. Temporary measures such as pheresis or hydrea (0.5 to 5g daily or more for up to 3 days) are allowed
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 3 year

SECONDARY OUTCOMES:
WT1 and MDR1 expression level change after 2 courses of chemotherapy with IA regimen or DA regimen in high-MDR1 expression AML patients. | 3 years

OTHER OUTCOMES:
Identify whether induction therapy with IA regimen has a higher remission quality with AML patients than that of DA regimen in high MDR1 expression AML patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, M.D, Study Chair — Department of Hematology, Nanfang Hospital, The Southern Medical University
Locations (1):
- Bing Xu, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Shi P, Zha J, Guo X, Chen F, Fan Z, Huang F, Meng F, Liu X, Feng R, Xu B. Idarubicin is superior to daunorubicin in remission induction of de novo acute myeloid leukemia patients with high MDR1 expression. Pharmacogenomics. 2013 Jan;14(1):17-23. doi: 10.2217/pgs.12.182. PMID 23252945
- See also: Nanfang Hospital, The Southern Medical University — http://www.nfyy.com/